CLINICAL TRIAL: NCT03428958
Title: A Phase Ib/II Open Label Study to Assess the Safety and Pharmacokinetics of NUC-3373, a Nucleotide Analogue, Given in Combination With Standard Agents Used in Colorectal Cancer Treatment
Brief Title: A Safety, Pharmacokinetic and Efficacy Study of NUC-3373 in Combination With Standard Agents Used in Colorectal Cancer Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NuCana plc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NuTide:302; 2017-002062-53 (EudraCT Number)
Record Dates: First submitted 2018-02-02; First posted 2018-02-12 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: Relapsed metastatic adenocarcinoma of colon/rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Leucovorin; Levoleucovorin; Oxaliplatin; Bevacizumab; Cetuximab; Panitumumab; Irinotecan

STUDY DESIGN:
Intervention Model Description: This is a three-part study of NUC-3373 administered by IV across two administration schedules, either as monotherapy or as part of various combinations with agents commonly used to treat CRC (LV, oxaliplatin, irinotecan, bevacizumab, cetuximab and panitumumab).
  Part 1 will determine if NUC-3373 should be administered with LV. Part 2 consists of a dose escalation phase, to assess the safety/tolerability of different doses of NUC-3373 in combination with either oxaliplatin (NUFOX) or irinotecan (NUFIRI), and an expansion phase, to assess weekly schedules of NUFOX and NUFIRI regimens selected in the escalation phase. Part 3 will assess the safety/efficacy of NUFOX and NUFIRI regimens administered in combination with bevacizumab, cetuximab or panitumumab.
  Additional patients may be enrolled in all parts to replace patients who withdraw prior to completing the 28-day safety evaluation period to complete the min number patients per cohort. Enrolment may be expanded at the DSMCs discretion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- NUC-3373 + leucovorin (LV) every other week (Experimental): Arm 1a: NUC-3373 administered IV followed by a 2-week washout period. The next dose of NUC-3373 administered in combination with LV at 400 mg/m2. All subsequent doses of NUC-3373 administered in combination with LV every 2 weeks in 28-day cycles.
  Interventions: Drug: NUC-3373 + leucovorin
- NUC-3373 every other week (Experimental): Arm 1b: LV 400 mg/m2 administered IV over 2 hours prior to NUC-3373 infusion followed by a 2-week washout period. Then, NUC-3373 administered IV every 2 weeks without LV in 28-day cycles.
  Interventions: Drug: NUC-3373
- NUC-3373 + leucovorin (LV) weekly (Experimental): Arm 1c: LV 400 mg/m2 administered IV over 2 hours followed by NUC-3373 administered IV weekly on Days 1, 8, 15 and 22 of 28-day cycles.
  Interventions: Drug: NUC-3373 + leucovorin
- NUC-3373 + leucovorin (LV); combination chemotherapy ineligible (Experimental): Arm 1d: LV 400 mg/m2 administered IV over 2 hours followed by NUC-3373 administered IV on Days 1, 8, 15 and 22 of 28-day cycles.
  Interventions: Drug: NUC-3373 + leucovorin
- NUC-3373 + oxaliplatin weekly (Experimental): Arm 2a: NUC-3373+LV (400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with oxaliplatin (85 mg/m2) administered on Days 1 and 15.
  Interventions: Drug: NUFOX
- NUC-3373 + irinotecan weekly (Experimental): Arm 2b: NUC-3373+LV (400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with irinotecan (180 mg/m2) on Days 1 and 15.
  Interventions: Drug: NUFIRI
- NUC-3373 + oxaliplatin (NUFOX) expansion (Experimental): Arm 2c: At the completion of Arm 2a, the recommended dose of NUC-3373 (+LV 400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with oxaliplatin (85 mg/m2) administered on Days 1 and 15.
  Interventions: Drug: NUFOX
- NUC-3373 + irinotecan (NUFIRI) expansion (Experimental): Arm 2d: At the completion of Arm 2b, the recommended dose of NUC-3373 (+LV 400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with irinotecan (180 mg/m2) on Days 1 and 15.
  Interventions: Drug: NUFIRI
- NUFOX + bevacizumab weekly (Experimental): Arm 3a: NUC-3373, LV and oxaliplatin at dose levels used in Arm 2a will be combined with bevacizumab. NUC-3373+LV will be administered weekly, oxaliplatin and bevacizumab will be administered every other week.
  Interventions: Drug: NUFOX + VEGF pathway inhibitor
- NUFOX + bevacizumab every other week (Experimental): Arm 3b: NUC-3373, LV and oxaliplatin at dose levels used in Arm 2a will be combined with bevacizumab. NUC-3373+LV+oxaliplatin+bevacizumab will be administered every other week.
  Interventions: Drug: NUFOX + VEGF pathway inhibitor
- NUFIRI + bevacizumab weekly (Experimental): Arm 3c: NUC-3373, LV and irinotecan at dose levels used in Arm 2b will be combined with bevacizumab. NUC-3373+LV will be administered weekly, irinotecan and bevacizumab will be administered every other week.
  Interventions: Drug: NUFIRI + VEGF pathway inhibitor
- NUFIRI + bevacizumab every other week (Experimental): Arm 3d: NUC-3373, LV and irinotecan at dose levels used in Arm 2b will be combined with bevacizumab. NUC-3373+LV+irinotecan+bevacizumab will be administered every other week.
  Interventions: Drug: NUFIRI + VEGF pathway inhibitor
- NUC-3373 + LV + bevacizumab; maintenance patients (Experimental): Arm 3e: NUC-3373+LV (400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with bevacizumab (administered every other week).
  Interventions: Drug: NUC-3373 + bevacizumab
- NUFOX + cetuximab (Experimental): Arm 3f: NUC-3373, LV and oxaliplatin at dose levels used in Arm 2a may be administered in subsequent cetuximab cohorts. NUC-3373+LV may be administered weekly or every other week, oxaliplatin will be administered every other week and cetuximab will be administered weekly.
  Interventions: Drug: NUFOX + EGFR inhibitor
- NUFIRI + cetuximab (Experimental): Arm 3g: NUC-3373, LV and irinotecan at dose levels used in Arm 2b may be administered in subsequent cetuximab cohorts. NUC-3373+LV may be administered weekly or every other week, irinotecan will be administered every other week and cetuximab will be administered weekly.
  Interventions: Drug: NUFIRI + EGFR inhibitor

INTERVENTIONS:
Drug: NUC-3373 + leucovorin — NUC-3373 + leucovorin
  Other Names: folinic acid; levoleucovorin; Nucleotide analogue
  Arms: NUC-3373 + leucovorin (LV) every other week; NUC-3373 + leucovorin (LV) weekly; NUC-3373 + leucovorin (LV); combination chemotherapy ineligible
Drug: NUC-3373 — NUC-3373
  Other Names: Nucleotide analogue
  Arms: NUC-3373 every other week
Drug: NUFOX — NUC-3373 + oxaliplatin
  Other Names: Eloxatin; Nucleotide analogue
  Arms: NUC-3373 + oxaliplatin (NUFOX) expansion; NUC-3373 + oxaliplatin weekly
Drug: NUFOX + VEGF pathway inhibitor — NUC-3373 + oxaliplatin + bevacizumab
  Other Names: Eloxatin; Avastin; Nucleotide analogue
  Arms: NUFOX + bevacizumab every other week; NUFOX + bevacizumab weekly
Drug: NUFOX + EGFR inhibitor — NUC-3373 + oxaliplatin + cetuximab/panitumumab
  Other Names: Eloxatin; Erbitux; Nucleotide analogue; Vectibix
  Arms: NUFOX + cetuximab
Drug: NUFIRI — NUC-3373 + irinotecan
  Other Names: Campto; Camptosar; Nucleotide analogue
  Arms: NUC-3373 + irinotecan (NUFIRI) expansion; NUC-3373 + irinotecan weekly
Drug: NUFIRI + VEGF pathway inhibitor — NUC-3373 + irinotecan + bevacizumab
  Other Names: Campto; Camptosar; Avastin; Nucleotide analogue
  Arms: NUFIRI + bevacizumab every other week; NUFIRI + bevacizumab weekly
Drug: NUFIRI + EGFR inhibitor — NUC-3373 + irinotecan + cetuximab/panitumumab
  Other Names: Campto; Camptosar; Erbitux; Nucleotide analogue; Vectibix
  Arms: NUFIRI + cetuximab
Drug: NUC-3373 + bevacizumab — NUC-3373 + bevacizumab
  Other Names: Nucleotide analogue; Avastin
  Arms: NUC-3373 + LV + bevacizumab; maintenance patients

SUMMARY:
This is a three-part study of NUC-3373 administered by intravenous (IV) infusion across two administration schedules, either as monotherapy or as part of various combinations with agents commonly used to treat CRC (leucovorin, oxaliplatin, irinotecan, bevacizumab, cetuximab and panitumumab). The primary objective is to identify a recommended dose and schedule for NUC-3373 when combined with these agents.

ELIGIBILITY:
Inclusion Criteria:

All patients

1. Provision of written informed consent
2. Have histological confirmation of CRC with evidence of locally advanced/unresectable or metastatic disease
3. Age ≥18 years
4. Life expectancy of ≥12 weeks
5. ECOG Performance status 0 or 1
6. Measurable disease as defined by RECIST v1.1
7. Known RAS and BRAF status. Patients with wild-type KRAS tumours who are to be enrolled to a cohort that does not contain an EGFR pathway inhibitor (Arms 2a, 2b, 2c, 2d, 3a, 3b, 3c, 3d and 3e) must have received prior treatment with an EGFR inhibitor, unless this was not standard of care according to relevant region-specific treatment recommendations. Patients with BRAF V600E mutant tumours should have received prior treatment with encorafenib in combination with an EGFR inhibitor, unless this was not standard of care according to relevant region-specific treatment recommendations
8. Adequate bone marrow function as defined by: ANC ≥1.5×10^9/L, platelet count ≥100×10^9/L (with no evidence of bleeding), and haemoglobin ≥9 g/dL
9. Adequate liver function as defined by serum total bilirubin ≤1.5×ULN, AST and ALT ≤2.5×ULN (or ≤5×ULN if liver metastases present)
10. Adequate renal function assessed as serum creatinine <1.5×ULN or glomerular filtration rate ≥50 mL/min. This criterion does not apply to Arm 1d.
11. Serum albumin ≥3 g/dL
12. For the cohort in which the patient will participate, there are no contra-indications to receiving the approved partner combination drugs
13. Ability to comply with protocol requirements
14. Female patients of child-bearing potential must have a negative serum pregnancy test within 7 days prior to the first study drug administration. This criterion does not apply to patients who have had a previous hysterectomy or bilateral oophorectomy. Male patients and female patients of child-bearing potential must agree to practice true abstinence or to use two highly effective forms of contraception, one of which must be a barrier method.
15. Patients must have been advised to take measures to avoid or minimise exposure to UV light for the duration of study participation and for a period of 4 weeks following the last dose of study medication
16. Male patients receiving oxaliplatin must have been offered advice on and/or sought counselling for conservation of sperm prior to the first dose of study medication

>3rd-line patients

1. Received at least two prior lines of therapy for locally advanced or metastatic CRC, including one fluoropyrimidine plus oxaliplatin and one fluoropyrimidine plus irinotecan containing regimen. Previous treatment with SoC regimens in combination with molecular targeted therapies is permitted and patients who received FOLFOXIRI-based regimens in 1st-/2nd-line settings may be included.
2. Patients due to receive NUFOX should be suitable for re-challenge with an oxaliplatin-based regimen
3. Patients due to receive NUFIRI should be suitable for re-challenge with an irinotecan-based therapy

2nd-/3rd-line patients

1. Received at least one but no more than two prior lines of fluoropyrimidine-containing therapy in combination with oxaliplatin and/or irinotecan for locally advanced or metastatic CRC. Previous treatment with SoC regimens in combination with molecular targeted therapies is permitted and patients who received FOLFOXIRI-based regimens in 1st-/2nd-line settings may be included. 3rd-line patients enrolled to Arms 2c and 2d must have received prior bevacizumab treatment, unless ineligible or unless bevacizumab was not standard of care according to relevant region-specific treatment recommendations
2. Patients in Part 2 due to receive NUFOX should be suitable for re-challenge with an oxaliplatin-based regimen
3. Patients in Part 2 due to receive NUFIRI should be suitable for re-challenge with an irinotecan-based regimen

Combination chemotherapy ineligible patients

1. May have received one prior fluoropyrimidine-containing regimen for locally advanced or metastatic CRC
2. Ineligible to receive combination therapy for locally advanced or metastatic CRC
3. Creatinine clearance >30mL/min

Rapid progressors

1. Received no more than two prior lines of fluoropyrimidine-containing therapy in combination with oxaliplatin and/or irinotecan for locally advanced or metastatic CRC. Previous treatment with SoC regimens in combination with molecular targeted therapies is permitted and patients who received FOLFOXIRI-based regimens in 1st-/2nd-line settings may be included.
2. Have had tumour progression ≤3 months of starting the last fluoropyrimidine-containing regimen
3. Patients due to receive NUFOX should be suitable for re-challenge with an oxaliplatin-based regimen
4. Patients due to receive NUFIRI should be suitable for re-challenge with an irinotecan-based regimen

2nd-line patients

1. Received one prior line of fluoropyrimidine-containing therapy in combination with oxaliplatin and/or irinotecan for locally advanced or metastatic CRC. Previous treatment with SoC regimens in combination with molecular targeted therapies is permitted and patients who received triplet chemotherapy based regimens is allowed.

Maintenance patients

1. Received at least 12 weeks of 1st-line SoC therapy for locally advanced or metastatic CRC and achieved at least stable disease
2. Eligible for maintenance therapy

Exclusion Criteria:

All patients

1. Prior history of hypersensitivity or current contra-indications to 5-FU or capecitabine
2. Prior history of hypersensitivity or current contra-indications to any of the combination agents required for the study arm to which the patient is assigned
3. History of allergic reactions attributed to the components of the NUC-3373 drug product formulation
4. Symptomatic CNS or leptomeningeal metastases
5. Symptomatic ascites, ascites currently requiring drainage procedures or ascites requiring drainage over the prior 3 months
6. Chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy [e.g. for bone pain]), immunotherapy or exposure to another investigational agent within 28 days (or five times half-life for a biological or molecular targeted agent or three times the half-life for an immunotherapy agent) of first receipt of study drug
7. Residual toxicities from prior chemotherapy or radiotherapy, which have not regressed to Grade ≤1 severity (CTCAE v5.0) except for alopecia. In cohorts not containing oxaliplatin, residual Grade 2 neuropathy is allowed.
8. History of another malignancy diagnosed within the past 5 years, with the exception of adequately treated non-melanoma skin cancer curatively treated carcinoma in situ of the cervix, surgically excised or potentially curatively treated ductal carcinoma in situ of the breast, or low grade prostate cancer or patients after prostatectomy not requiring treatment. Patients with previous invasive cancers are eligible if treatment was completed more than 3 years prior to initiating the current study treatment and there is no evidence of recurrence.
9. Presence of active bacterial or viral infection (including SARS-CoV-2, Herpes Zoster or chicken pox), known HIV positive or known active hepatitis B or C
10. Presence of any uncontrolled concurrent serious illness, medical condition or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with their participation in the study, or with the interpretation of the results
11. Any condition (e.g. known or suspected poor compliance, psychological instability, geographical location) that, in the judgment of the Investigator, may affect the patient's ability to sign the informed consent and undergo study procedures
12. Currently pregnant, lactating or breastfeeding
13. QTc interval >450 milliseconds for males and >470 milliseconds for females
14. Required concomitant use of drugs known to prolong QT/QTc interval
15. Required concomitant use of strong CYP3A4 inducers or strong CYP3A4 inhibitors, or use of strong CYP3A4 inducers within 2 weeks of first receipt of study drug or use of strong CYP3A4 inhibitors within 1 week of first receipt of study drug
16. For patients receiving irinotecan: Use of strong UGT1A1 inhibitors within 1 week of first receipt of study drug
17. Has received a live vaccination within four weeks of first planned dose of study medication
18. Known DPD or TYMP mutations associated with toxicity to fluoropyrimidines
19. Use of warfarin and other types of long acting anti-coagulants is prohibited within 4 weeks of the first dose of study treatment

Patients receiving bevacizumab

1. Patients with a history of haemoptysis (≥1/2 tsp of red blood)
2. Wound healing complications or surgery within 28 days of starting bevacizumab
3. Severe chronic wounds, ulcers or bone fracture
4. Arterial thromboembolic events or haemorrhage within 6 months prior to study entry (except for tumour bleeding surgically treated by tumour resection)
5. Bleeding diatheses or coagulopathy
6. Receiving full-dose anti-coagulation treatment
7. Uncontrolled hypertension
8. Clinically significant coronary heart disease or myocardial infarction within the last 12 months or high risk of uncontrolled arrhythmia
9. Severe proteinuria
10. Acute or subacute ileus, chronic inflammatory bowel disease or chronic diarrhoea
11. Any contraindications present in the bevacizumab Prescribing Information

Patients receiving cetuximab or panitumumab

1. Clinically significant coronary heart disease or myocardial infarction within the last 12 months or high risk of uncontrolled arrhythmia
2. Acute or subacute ileus, chronic inflammatory bowel disease or chronic diarrhoea
3. Hypomagnesaemia or hypokalaemia not controlled by oral therapy
4. Any contraindications present in the cetuximab or panitumumab Prescribing Information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Oelmann, MD PhD, Study Director — NuCana plc
Locations (10):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Seattle Cancer Center, Seattle, Washington
  - Compass Oncology, Vancouver, Washington
- Hopital Franco-Britannique, Levallois-Perret, France
- United Kingdom (3):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 111 patients were recruited between July 2018 and June 2023.
Pre-assignment Details: No participants were recruited in Arms 1d, 2c, 2d, 3b, 3d, 3e, 3f, and 3g
Groups:
- NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly: Arm 1c: LV 400 mg/m2 administered IV over 2 hours followed by NUC-3373 1500 mg/m2 administered IV weekly on Days 1, 8, 15 and 22 of 28-day cycles.
  NUC-3373 + leucovorin: NUC-3373 + leucovorin
- NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly: Arm 1c: LV 400 mg/m2 administered IV over 2 hours followed by NUC-3373 2500 mg/m2 administered IV weekly on Days 1, 8, 15 and 22 of 28-day cycles.
  NUC-3373 + leucovorin: NUC-3373 + leucovorin
- NUC-3373 + Irinotecan Weekly (PK Sub-study): Arm 2b (PK sub-study): NUC-3373+LV (400 mg/m2) administered weekly on Days 1, 8, 15 and 22 of 28-day cycles in combination with irinotecan (180 mg/m2) on Days 1 and 15.
  NUFIRI: NUC-3373 + irinotecan
Period: Overall Study
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Leucovorin (LV); Combination Chemotherapy Ineligible | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUC-3373 + Oxaliplatin (NUFOX) Expansion | NUC-3373 + Irinotecan (NUFIRI) Expansion | NUFOX + Bevacizumab Weekly | NUFOX + Bevacizumab Every Other Week | NUFIRI + Bevacizumab Weekly | NUFIRI + Bevacizumab Every Other Week | NUC-3373 + LV + Bevacizumab; Maintenance Patients | NUFOX + Cetuximab | NUFIRI + Cetuximab
Started | 11 | 11 | 12 | 6 | 0 | 23 | 25 | 9 | 0 | 0 | 5 | 0 | 9 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 11 | 12 | 6 | 0 | 23 | 25 | 9 | 0 | 0 | 5 | 0 | 9 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 2 | 3 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progression per RECIST | 6 | 6 | 7 | 4 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0 | 0 | 7 | 9 | 6 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician/Sponsor Decision | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients recruited to Arms 1d, 2c, 3b, 3d, 3e, 3f, and 3g.
Groups:
- Total: Total of all reporting groups
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Leucovorin (LV); Combination Chemotherapy Ineligible | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUC-3373 + Oxaliplatin (NUFOX) Expansion | NUC-3373 + Irinotecan (NUFIRI) Expansion | NUFOX + Bevacizumab Weekly | NUFOX + Bevacizumab Every Other Week | NUFIRI + Bevacizumab Weekly | NUFIRI + Bevacizumab Every Other Week | NUC-3373 + LV + Bevacizumab; Maintenance Patients | NUFOX + Cetuximab | NUFIRI + Cetuximab | Total
Number analyzed (Participants) | 11 | 11 | 12 | 6 | 0 | 23 | 25 | 9 | 0 | 0 | 5 | 0 | 9 | 0 | 0 | 0 | 0 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (13.2) | 59.1 (9.3) | 55.4 (10.2) | 56.0 (11.0) |  | 58.3 (10.0) | 56.7 (10.1) | 55.3 (10) |  |  | 65 (5.9) |  | 54.3 (14.2) |  |  |  |  | 57 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 4 |  | 12 | 10 | 7 |  |  | 2 |  | 3 |  |  |  |  | 51
  Male | 7 | 6 | 8 | 2 |  | 11 | 15 | 2 |  |  | 3 |  | 6 |  |  |  |  | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 |  | 1 | 1 | 1 |  |  | 0 |  | 0 |  |  |  |  | 4
  Not Hispanic or Latino | 11 | 11 | 10 | 6 |  | 21 | 21 | 8 |  |  | 4 |  | 7 |  |  |  |  | 99
  Unknown or Not Reported | 0 | 0 | 1 | 0 |  | 1 | 3 | 0 |  |  | 1 |  | 2 |  |  |  |  | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 |  | 0 | 0 | 0 |  |  | 0 |  | 0 |  |  |  |  | 1
  Asian | 0 | 0 | 1 | 0 |  | 1 | 2 | 1 |  |  | 1 |  | 1 |  |  |  |  | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 1 | 0 | 0 |  |  | 0 |  | 0 |  |  |  |  | 1
  Black or African American | 1 | 1 | 0 | 0 |  | 0 | 2 | 0 |  |  | 0 |  | 1 |  |  |  |  | 5
  White | 10 | 10 | 10 | 5 |  | 20 | 19 | 8 |  |  | 4 |  | 7 |  |  |  |  | 93
  More than one race | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 |  |  | 0 |  | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 |  | 1 | 2 | 0 |  |  | 0 |  | 0 |  |  |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Tumour Size
Description: Efficacy (per RECIST v 1.1): defined as the best percentage change from baseline in tumour size (mm)
Time Frame: Assessed every 8 weeks following Day 1 until the end of study (up to 25 months)
Population: Evaluable for Response (EFR): Patients with measurable disease at baseline who received at least two cycles of study treatment (receiving at least 75% of the planned doses over the two cycles) and had a post-treatment objective disease assessment. Data are only available for patients in the EFR set who did not have a best response of progressive disease and who had evaluable post-dose target lesion data. All patients in Arm 1a had a best response of either progressive disease or non-evaluable.
Measure: Median (Full Range); unit: Percent change
Groups:
- NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly; NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly: Arm 1c: LV 400 mg/m2 administered IV over 2 hours followed by NUC-3373 administered IV weekly on Days 1, 8, 15 and 22 of 28-day cycles.
  NUC-3373 + leucovorin: NUC-3373 + leucovorin
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 0 | 4 | 5 | 2 | 8 | 9 | 2 | 4 | 8
Percent change |  | 8.3 [-15 to 20] | 2.9 [-28 to 15] | 3.2 [-3 to 9] | 2.3 [-19 to 10] | 7.9 [-12 to 21] | 2.8 [-2 to 8] | -13.9 [-18 to -12] | -11.1 [-26 to 5]

2. Primary Outcome: Disease Control Rate (DCR)
Description: Efficacy (per RECIST v 1.1): defined as the proportion of patients achieving confirmed response (CR and PR) or stable disease (SD) as the best overall response
Time Frame: Assessed every 8 weeks following Day 1 until the end of study (up to 25 months)
Population: Evaluable for Response (EFR): Patients with measurable disease at baseline who received at least two cycles of study treatment (receiving at least 75% of the planned doses over the two cycles) and had a post-treatment objective disease assessment. Data are only available for patients in the EFR set achieving confirmed response (CR and PR) or stable disease (SD) as the best overall response.
Measure: Number; unit: percentage of patients
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 3 | 7 | 8 | 4 | 15 | 14 | 6 | 5 | 9
percentage of patients | 0 | 42.9 | 62.5 | 50 | 46.7 | 42.9 | 33.3 | 80.0 | 88.9

3. Primary Outcome: Duration of Stable Disease (DoSD)
Description: Efficacy (per RECIST v 1.1): defined as the time from the time measurement criteria are first met for SD until the first date that recurrence or progressive disease (PD) is objectively documented
Time Frame: Assessed every 8 weeks following Day 1 until the end of study (up to 25 months)
Population: Evaluable for Response (EFR): Patients with measurable disease at baseline who received at least two cycles of study treatment (receiving at least 75% of the planned doses over the two cycles) and had a post-treatment objective disease assessment. Data are only available for patients in the EFR set who did not have a best response of progressive disease and who had evaluable post-dose target lesion data and had Stable Disease.
Measure: Median (Full Range); unit: months
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 0 | 3 | 5 | 2 | 7 | 6 | 2 | 4 | 8
months |  | 1.9 [1.9 to 4.8] | 2.6 [0.03 to 3.3] | 1.9 [1.9 to 1.9] | 3.7 [0.03 to 4.4] | 3.2 [2.0 to 8.6] | 2.3 [2.0 to 2.5] | 6.5 [5.3 to 7.9] | 4.6 [0.2 to 13.2]

4. Primary Outcome: Progression Free Survival (PFS)
Description: Efficacy (per RECIST v 1.1): defined as the time from first dose of study treatment until the date of objective disease progression or death
Time Frame: Assessed every 8 weeks following Day 1 until the end of study (up to 25 months)
Population: Patients who received at least one dose of NUC-3373
Measure: Median (Full Range); unit: months
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 10 | 11 | 11 | 6 | 23 | 23 | 8 | 5 | 9
months | 1.7 [0.03 to 2.1] | 2.3 [0.03 to 4.2] | 2.9 [0.03 to 5.0] | 1.8 [0.03 to 3.6] | 2.5 [0.03 to 6.1] | 3.6 [0.03 to 6.5] | 2.0 [0.03 to 4.1] | 7.7 [2.3 to 9.8] | 5.5 [1.9 to 15.0]

5. Primary Outcome: Overall Survival (OS)
Description: Efficacy: defined as the time from randomization until the date of death from any cause
Time Frame: From the date of randomization until the date of death from any cause, until the end of study (up to 25 months)]
Population: Full Analysis Set: All randomised patients
Measure: Median (Full Range); unit: months
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 11 | 11 | 12 | 6 | 23 | 25 | 9 | 5 | 9
months | 1.9 [0.9 to 3.3] | 3.0 [1.5 to 7.7] | 3.6 [0.8 to 8.0] | 3.6 [1.3 to 5.5] | 3.4 [0.4 to 24.5] | 3.2 [0.5 to 19.1] | 7.3 [1.4 to 13.6] | 14.2 [9.4 to 16.9] | 12.8 [3.2 to 18.2]

6. Primary Outcome: Best Overall Response
Description: Best overall response to study treatment according to RECIST v1.1
Time Frame: Assessed every 8 weeks from Day 1 until the end of study (up to 25 months)
Population: Evaluable for Response (EFR): Patients with measurable disease at baseline who received at least two cycles of study treatment (receiving at least 75% of the planned doses over the two cycles) and had a post-treatment objective disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
Number analyzed (Participants) | 3 | 7 | 8 | 4 | 15 | 14 | 6 | 5 | 9
percentage of participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 42.9 | 62.5 | 50 | 46.7 | 42.9 | 33.3 | 80.0 | 88.9
  Progressive Disease | 100.0 | 42.9 | 37.5 | 50.0 | 46.7 | 42.9 | 66.7 | 20.0 | 11.1
  Not Evaluable | 0 | 14.3 | 0 | 0 | 6.7 | 14.3 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Each patient was assessed for serious and other (non-serious) adverse events from the date of consent until 30 days after the last dose of study treatment, up to 25 months. Each patient was assessed for all-cause mortality from the date of randomization until the date of death from any cause, up to 25 months.
Description: All-Cause Mortality was assessed for the Full Analysis Set.
  Serious Adverse Events and/or Other (Not Including Serious) Adverse Events were assessed for the Safety Population (all participants that received at least one dose of NUC-3373).
Arm/Group | NUC-3373 + Leucovorin (LV) Every Other Week | NUC-3373 Every Other Week | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly | NUC-3373 + Oxaliplatin Weekly | NUC-3373 + Irinotecan Weekly | NUC-3373 + Irinotecan Weekly (PK Sub-study) | NUFOX + Bevacizumab Weekly | NUFIRI + Bevacizumab Weekly
All-Cause Mortality (participants affected / at risk) | 3/11 | 4/11 | 1/12 | 0/6 | 11/23 | 11/25 | 6/9 | 3/5 | 4/9
Serious Adverse Events (participants affected / at risk) | 6/10 | 2/11 | 3/11 | 2/6 | 11/23 | 8/23 | 2/8 | 4/5 | 4/9
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11 | 11/11 | 6/6 | 23/23 | 23/23 | 8/8 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NUC-3373 + Leucovorin (LV) Every Other Week (N=10) | NUC-3373 Every Other Week (N=11) | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly (N=11) | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly (N=6) | NUC-3373 + Oxaliplatin Weekly (N=23) | NUC-3373 + Irinotecan Weekly (N=23) | NUC-3373 + Irinotecan Weekly (PK Sub-study) (N=8) | NUFOX + Bevacizumab Weekly (N=5) | NUFIRI + Bevacizumab Weekly (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NUC-3373 + Leucovorin (LV) Every Other Week (N=10) | NUC-3373 Every Other Week (N=11) | NUC-3373 (1500 mg/m2) + Leucovorin (LV) Weekly (N=11) | NUC-3373 (2500 mg/m2) + Leucovorin (LV) Weekly (N=6) | NUC-3373 + Oxaliplatin Weekly (N=23) | NUC-3373 + Irinotecan Weekly (N=23) | NUC-3373 + Irinotecan Weekly (PK Sub-study) (N=8) | NUFOX + Bevacizumab Weekly (N=5) | NUFIRI + Bevacizumab Weekly (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 | 4 | 1 | 10 | 10 | 3 | 3 | 3
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 1 | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 1 | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 5 (7) | 7 (8) | 4 (5) | 2 (2) | 4 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 8 (13) | 4 (7) | 4 (5) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (6) | 1 (11) | 10 (27) | 15 (21) | 4 (4) | 4 (11) | 8 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 7 (9) | 4 (18) | 13 (24) | 13 (20) | 4 (8) | 5 (12) | 5 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 8 (11) | 4 (10) | 13 (26) | 8 (9) | 2 (2) | 4 (8) | 5 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 2 (2) | 1 (2) | 5 (13) | 15 (24) | 8 (15) | 8 (8) | 4 (4) | 6 (9)
Feeling hot (General disorders) | 2 (4) | 2 (2) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 2 (4) | 1 (5) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sweating fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pruritus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (4) | 1 (5) | 6 (9) | 2 (8) | 1 (1) | 0 (0) | 5 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 5 (8) | 4 (6) | 1 (1) | 0 (0) | 5 (15)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 9 (9) | 6 (7) | 2 (2) | 2 (3) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (4) | 2 (2) | 2 (3) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (4) | 3 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (8) | 4 (5) | 2 (2) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (8) | 2 (2) | 1 (1) | 2 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 4 (7) | 1 (2) | 1 (1) | 3 (5) | 4 (6) | 2 (4) | 0 (0) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 3 (6) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03428958/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT03428958/SAP_001.pdf